CLINICAL TRIAL: NCT00135447
Title: A Phase IV, Multicenter, Cross-sectional Study to Evaluate the I50L Substitution Among Subjects Experiencing Virologic Failure on a HAART Regimen Containing Atazanavir (ATV)
Brief Title: A Study of Prevalence of the I50L Mutation When ATV Treated Patients Fail the Regimen
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Other Study IDs: AI424-128
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: HIV Infections
Keywords: HIV/AIDS; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A

SUMMARY:
The purpose of this study is to find out the frequency of the I50L substitution among patients experiencing treatment failure on an atazanavir-containing regimen.

ELIGIBILITY:
Inclusion Criteria:

* Atazanavir - containing antiretroviral regimen
* Confirmed virologic failure defined as either:

  1. HIV RNA by PCR greater than or equal to 1000 copies/mL after achieving a value of <400 copies/mL on at least 2 consecutive measurements or
  2. HIV RNA greater than or equal to 1000 copies/mL after 24 weeks of continuous therapy
* At least 18 years old

Exclusion Criteria:

* Unable to give informed consent
* Prisoners or subjects involuntarily incarcerated for treatment of psychiatric or physical illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV infected patients failing HAART regimen
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2004-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (84):
- United States (84):
  - Local Institution, Phoenix, Arizona
  - Vista Medical Partners, Beverly Hills, California
  - AIDS Healthcare Foundation, Beverly Hills, California
  - AltaMed Health Services Corporation, Los Angeles, California
  - Kaiser Permanente, Los Angeles, California
  - Synergy Hematology and Oncology Medical Associates, Los Angeles, California
  - Orange Coast Medical Group, Newport Beach, California
  - Alameda County Medical Center, Oakland, California
  - East Bay AIDS Center, Oakland, California
  - Desert Medical Group, Palm Springs, California
  - Martin M. Mass, MD, San Francisco, California
  - Wellspring Medical Group, San Francisco, California
  - San Mateo Medical Center, San Mateo, California
  - Stanford University Medical Center, Stanford, California
  - Denver Public Health, Denver, Colorado
  - Local Institution, Denver, Colorado
  - Dupont Circle Physicians Group, P.C., Washington D.C., District of Columbia
  - South Florida Clinical Research, Atlantis, Florida
  - Daniel A. Warner, MD, PA, Daytona Beach, Florida
  - Gary J. Richmond, MD, PA, Fort Lauderdale, Florida
  - Biogenomx Research Institute, LLC/CHC1-AP, Hollywood, Florida
  - AIDS Healthcare Foundation, Jacksonville, Florida
  - Steinhart Medical Associates, Miami, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Care Resource, Inc., Miami, Florida
  - Albert Canas MD, PA, Miami Beach, Florida
  - Associates in Infectious Diseases, Port Saint Lucie, Florida
  - Health Positive, Safety Harbor, Florida
  - Bach & Godofsky, MD, PA, Sarasota, Florida
  - Edward W. Braun, MD PA, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Grady Ponce de Leon Infectious Disease Clinic, Atlanta, Georgia
  - Atlanta ID Group, Atlanta, Georgia
  - Infectious Disease Solutions, Atlanta, Georgia
  - Infectious Disease Group of Atlanta, Atlanta, Georgia
  - Family Healthcare of Atlanta, PC, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Investious Diseases Associates, Riverdale, Georgia
  - Southern Illinois University of Medicine, Springfield, Illinois
  - University of Iowa Healthcare, Iowa City, Iowa
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Chase Brexton Health Services, Baltimore, Maryland
  - University of Maryland, Institute of Human Virology, Baltimore, Maryland
  - St. Agnes Health Care, Inc., Baltimore, Maryland
  - Calvert Internal Medicine Group, Prince Frederick, Maryland
  - Tufts New England Medical Center, Boston, Massachusetts
  - Fenway Community Health, Boston, Massachusetts
  - The Research Institute, Springfield, Massachusetts
  - Be Well Medical Center, Berkley, Michigan
  - Michaigan State Adult Medicine Clinic, Lansing, Michigan
  - Charles P. Craig, M.D., P.C., Ypsilanti, Michigan
  - Central West Clinical Research, Inc., St Louis, Missouri
  - Garden State Infectious Disease Associates, Voorhees Township, New Jersey
  - Philip S. Smith, MD, Cornwall-on-Hudson, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Beth Israel Medical Center, New York, New York
  - Ricky K. Hsu, MD, PC, New York, New York
  - Ronald Grossman, MD, New York, New York
  - AIDS Community Research Initiative of America, New York, New York
  - James Jones, MD, New York, New York
  - New York Medical College, Valhalla, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Local Institution, Charlotte, North Carolina
  - Fairgrove Primary Health, Hickory, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Metro Heath Medical Center, Cleveland, Ohio
  - The University of Toledo, Toledo, Ohio
  - The Research and Education Group, Portland, Oregon
  - Kaiser Permanente Northwest Region, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Univeristy Speciality Clinics, Columbia, South Carolina
  - Greenville Hospital System, Greenville, South Carolina
  - Nicholaos C. Bellos, MD, Dallas, Texas
  - Amelia Court HIV Research, Dallas, Texas
  - Planned Parenthood Center of El Paso, El Paso, Texas
  - Tarrant Country Infectious Disease Associates, Fort Worth, Texas
  - Valley AIDS Council, Harlingen, Texas
  - Therapeutic Concepts, P.A., Houston, Texas
  - Diversified Medical Pratices, PA, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Medical Associates of Central Virginia, Lynchburg, Virginia
  - Richmond AIDS Consortium, Richmond, Virginia
  - Daniel R. Coulston, MD, Spokane, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin